CLINICAL TRIAL: NCT06404645
Title: A Clinical Prospective Observational Study of Near Infrared Spectroscopy to Detect Subcranial Hematoma
Acronym: NIRS-DETECT
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2024-054-B
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Near-infrared spectroscopy detection — Cranial CT confirm intracranial haematoma. Then the near-infrared spectroscopy device to collect date by red sensor probe in the corresponding position on the scalp and blue sensor probe on the opposite side of the hematoma. Collect data for 10 minutes.

SUMMARY:
This trial is a clinical prospective observational study. Cases meeting the entry criteria undergo near-infrared spectroscopy(NIRS）detection. Data collection mainly includes hematoma thickness on cranial CT, and bilateral NIRS data.This trial tries to explore the reliability and accuracy of NIRS detection of subcranial hematoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years old
2. Unilateral subcranial hemorrhage confirmed by cranial CT

Exclusion Criteria:

1. Bilateral subcranial hemorrhage
2. Intracranial pneumoperitoneum in the location of the hemorrhage on cranial CT
3. Obvious skull fracture in the location of hemorrhage on cranial CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergo cranial CT that reveal a unilateral intracranial hemorrhage. Once meeting the inclusion and exclusion criteria, patients sign an informed consent and then undergo NIRS test.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
NIRS data1 | 3 months
  NIRS data of bleeding side and the opposite side

SECONDARY OUTCOMES:
NIRS data2 | 3 months
  relationship between NIRS data and thickness of haematoma

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Feng, Study Chair — RenJi Hospital
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No